CLINICAL TRIAL: NCT02306967
Title: Fluorescent Visualization in Early Oral Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Terry Fox Research Institute (Other)
Responsible Party: Principal Investigator, Joseph C. Dort, Professor of Surgery, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCENT004
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Oral Squamous Cell Carcinoma or Severe Dysplasia
Keywords: oral cancer; oral dysplasia
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Standard Resection (Active Comparator): Oral resection will be guided by usual practice. This involves identifying the tumour with white light and then marking surgical margins and resection the primary cancer.
  Interventions: Procedure: resection of oral cancer
- FV Guided Resection (Experimental): The oral resection will be guided by fluorescent visualization (FV).
  Interventions: Procedure: resection of oral cancer

INTERVENTIONS:
Procedure: resection of oral cancer — Oral cancer will be resected.
Procedure: resection of oral cancer — Oral cancer will be resected

SUMMARY:
Studies from Vancouver show that fluorescent visualization (FV) is a useful method of controlling surgical margins. This early finding will now be confirmed in a national randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven invasive oral cancer or severe dysplasia / Cis
* invasive cancer must be T1 or T2
* no prior history of oral cancer / treatment of oral cancer

Exclusion Criteria:

* prior history of oral cancer
* unable to provide informed consent
* lesion not able to be completely visualized by FV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
disease specific survival | 5 years
  disease specific 5 year survival

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada